CLINICAL TRIAL: NCT01255371
Title: A Multicenter Phase III Trial of Second-line Antiretroviral Treatment Strategies in African Adults (Tanzania Ans South Africa) Using Atazanavir or Lopinavir/Ritonavir
Brief Title: A Multicentre Trial of Second-line Antiretroviral Treatment Strategies in African Adults Using Atazanavir or Lopinavir/Ritonavir
Acronym: ALISA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: drug procurement issues
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Ludwig-Maximilians - University of Munich (Other); Institute of Tropical Medicine, Belgium (Other); Institut de Recherche pour le Developpement (Other Government); Swiss National Science Foundation (Other); University of Limpopo (Other); NIMR-Mbeya Medical Research Program (MMRP)/ Mbeya Referral Hospital, Tanzania (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12221 ALISA; IP.07.33011.004 (Other Grant/Funding Number: EDCTP)
Record Dates: First submitted 2010-11-29; First posted 2010-12-07 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: HIV
Keywords: HIV; Second line antiretroviral treatment; Sub saharian Africa; Generic
MeSH Terms: interventions — Lopinavir; Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A : Lopinavir (Active Comparator): Emtricitabine/tenofovir :
  * TDF300mg.FTC200mg (Fixed Dose Combination)
  * 1 tablet per day
  Lopinavir/ritonavir :
  * LPV200mg/RTV50mg
  * 2 tablets twice a day
  Interventions: Drug: Lopinavir
- Arm B : Atazanavir (Experimental): Lamivudine/tenofovir :
  * 3TC300mg/TDF300mg (Fixed Dose Combination)
  * 1 tablet per day
  Atazanavir/ritonavir :
  * ATV300mg/RTV100mg
  * 2 tablets once a day
  Interventions: Drug: Atazanavir

INTERVENTIONS:
Drug: Lopinavir — Evaluation of second line antiretroviral regimen including boosted lopinavir
  Arms: Arm A : Lopinavir
Drug: Atazanavir — Evaluation of second line antiretroviral regimen including boosted atazanavir
  Arms: Arm B : Atazanavir

SUMMARY:
In the well recognized context of HIV infection chronicity, it is now crucial to identify and evaluate effective, well tolerated and affordable second line regimen in resources limited countries where patients often change treatment after a long period of viral replication while on first line regimen.

This multicentre international, randomized, non-blinded phase III trial aim to demonstrate the non-inferiority of a generic lamivudine-tenofovir-atazanavir/ritonavir regimen (daily intake) as compared to a standard emtricitabine-tenofovir-lopinavir/ritonavir (twice daily intake)regimen for second line HIV-1 treatment. by stratifying on the viral load level (between 1000 and 5000 copies/mL versus > 5000 copies/mL) at inclusion, this trial will also allow to evaluate the optimum moment for instituting the second-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and above
* out patient
* documented HIV-1 infection
* first line treatment failure:

  * after first-line antiretroviral treatment with a combination including a non-nucleoside reverse transcriptase inhibitor and two nucleoside reverse transcriptase inhibitors
  * two measurements of plasma HIV RNA levels > 1000 copies/mL after at least 6 months of uninterrupted treatment or without any major modification
* satisfactory compliance (>80%) to 1st line antiretroviral treatment
* signed informed consent
* agreement for contraception for women of childbearing age

Exclusion Criteria:

* HIV-2 infection or HIV-1/HIV-2 coinfection
* uncontrolled, ongoing opportunistic infection or of any severe or progressive disease including active TB
* first line antiretroviral treatment with a protease inhibitor or tenofovir
* ongoing treatment with rifampicin
* severe hepatic insufficiency (PT < 50%)
* ALT < 3 times the upper limit of normal
* creatinine clearance calculated by Cockcroft's formula < 50 mL/min
* Hb <=8 g/dL; platelets < 50,000 cells/mm3; neutrophils < 500 cells/mm3
* pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Virological response | 48 weeks
  Proportion of patients with plasma HIV RNA < 50 copies/mL

SECONDARY OUTCOMES:
Virological response | 12 and 24 weeks
  Proportion of patients with plasma HIV RNA < 400 copies/mL
Viral resistance | 12, 24 and 48 weeks
  Incidence of resistance mutations after treatment failure (HIV RNA < 1000 copies/mL)
Clinical course of HIV infection | Up to 48 weeks
  Mortality, occurence of clinical events stage 3 or 4 (WHO classification), immune reconstitution sundrome, non-AIDS clinical events including bacterial infections
Tolerance assessment | 24 and 48 weeks
  Proportion of adverse events related to antiretroviral treatment, proportion of treatement discontinuations due to antiretroviral side effect, variation of biological parameters and metabolic markers between second line antiretroviral initiation and 24/48 weeks.
Adherence assessment | At each protocol visit : week 2, 4, 12, 24, 36 and 48
  Measurement of pills consumption at each visit, face-to-face questionnaire with the pharmacist
Hepatitis B evaluation | At entry
  Prevalence of HBs AG, HBe Ag, HBV viremia, and HBV asociated drug resistance mutations at baseline
Immunologic response | 24 and 48 weeks
  Variation of circulating total and CD4+ lymphocyte count between second line treatment initiation and 24 weeks/48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Delaporte, Principal Investigator — Institut de Recherche pour le Developpement; Issakwisa Mwakyula, Principal Investigator — NIMR-Mbeya Medical Research Program-Mbeya Referral Hospital, Tanzania; Mzileni O Mogiyana, Principal Investigator — University of Limpopo; Alexandra Calmy, Principal Investigator — University of Geneva, Switzerland
Locations (2):
- Tshepang clinic, Limpopo University, Pretoria, South Africa
- NIMR-Mbeya Medical Research Program-Mbeya Referral Hospital, Mbeya, Tanzania